CLINICAL TRIAL: NCT04849767
Title: Trans&VIH: National Survey About Trajectory and Life Conditions of HIV Trans People in France
Brief Title: National Survey About Trajectory and Life Conditions of HIV Trans People in France
Acronym: Trans&VIH
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 14056 TRANS&VIH; 20-694 (Other: The Inserm Ethics Evaluation Committee IRB00003888)
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2021-04

CONDITIONS: HIV Seropositivity
Keywords: Transgender; Community-based research; Mixt methods
MeSH Terms: conditions — HIV Seropositivity | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transgender people living with HIV: Transgender person Living with HIV Followed in clinical service
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire about socio-behavioral items and conditions of vulnerability. interview with female to male transgender person will be about life conditions, trajectory of the medical transition from female to male and actual medical following of the transition, migration trajectory and condition of HIV acquisition.
  Other Names: interview

SUMMARY:
TRANS&VIH is a national survey that will explore condition of vulnerability and trajectory of transgender people living with HIV. To fulfill this purpose, clinical data from medical registry and socio-behavioral information collected through questionnaire, will help to explore this questions about vulnerability and condition of transgender people living with HIV.

DETAILED DESCRIPTION:
In France, transgender still a taboo subject, and is poorly documented. There are no precise data on the number of transgender people in France or on their socio-demographic characteristics. The absence of such data reinforces their invisibility in social life and contributes to their stigmatization. Transgender people faces many social barriers in our society. These barriers accumulate in HIV seropositive transgender people (TRHIV), and most likely increase the burden of HIV infection. The main objective of ANRS TRANS&VIH - the community-based research study presented here - is to identify personal and social situations of vulnerability for TRHIV in France, the obstacles for receiving medical care, and their healthcare needs.

ANRS TRANS&VIH is an ongoing national, exhaustive, cross-sectional survey of all TRHIV currently followed up in HIV services in France. It is a mixed-methods study, the quantitative and qualitative components includ TRHIV women and men, respectively. Socio-behavioral and medical data are collected (start date January 2021) by community-based interviewers in participating hospital-based HIV structures in order to explore patient care pathways and living conditions of the TRHIV population with regard to transitioning and HIV. This is the first study in France to collect such data. The statistical techniques used for the data analyses will reflect the study's objectives and will be adapted to the type of data collection used: cross-sectional (questionnaires) and longitudinal (life history). Several types of analyses will be performed, including: (i) a description of the individual characteristics of transgender female TRHIV; (ii) comparative analyses between different groups of stakeholders (e.g., differences between the Ile de France region (which covers Paris and the surrounding area) and other regions); (iii) analysis of life and HIV trajectories; (iv) structural analyses using structural data collected for participating HIV structures (v) qualitative analysis of data from interviews with participating TRHIV men.

ANRS TRANS&VIH results will be used to make recommendations to health authorities to ensure that a comprehensive healthcare package will be offered to TRHIV which takes into account this population's specific background and problems.

ELIGIBILITY:
Inclusion Criteria:

* transgender woman or transgender man
* living with HIV
* followed in hospitals in metropolitan France and the country's overseas territories

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-define as transgender, or who present themselves with a gender different from the one they were assigned at birth (transgender woman or transgender man)
Study Population: People who self-define as transgender, or who present themselves with a gender different from the one they were assigned at birth (transgender woman or transgender man), living with HIV (TRHIV), and followed in hospitals in metropolitan France and the country's overseas territories.
  TRHIV frequenting hospital-based HIV services in France. In 2018, an exploratory survey in 258 such hospital services, allowed the estimation of the study population: 852 TRHIV women and 5 TRHIV men. Given the small size of the active patient file, we decided to survey all the TRHIV who agreed to participate in ANRS Trans & HIV, in order to highlight possible disparities in HIV and transition care.
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Statistical analyses of trends in the personal and social situations of vulnerability in TRHIV | 12 months
  Through statistical analyses of some questionnaire items, we will highlight the situations of vulnerability of transgender people.
Statistical analyses of trends in obstacles that TRHV encounter in terms of medical care and their healthcare needs | 12 months
  The results, of the analyses of questionnaire data, will point trends in the medical needs of the study population and the factors that hamper the satisfiction of these needs.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno SPIRE, Dr, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- INSERM, Marseille, France

REFERENCES:
- [Derived] Van Huizen R, Annequin M, Mora M, Faye A, Fiorentino M, Bourrelly M, Maradan G, Berenger C, Michard F, Yazdanpanah Y, Freire Maresca A, Rouveix E, Cuenot L, Balhan L, Costa M, Michels D, Blanquart L, Rincon G, Protiere C, Spire B; ANRS-Trans&HIV study group. Socioeconomic marginalization, social exclusion, and engagement in transactional sex among transgender women living with HIV: the role of multidimensional gender affirmation. AIDS Care. 2025 Dec;37(12):2174-2191. doi: 10.1080/09540121.2025.2560094. Epub 2025 Sep 29. PMID 41024590
- [Derived] Mora M, Rincon G, Bourrelly M, Maradan G, Freire Maresca A, Michard F, Rouveix E, Pannetier J, Leriche D, Alain T, Yazdanpanah Y, Michels D, Spire B. Living conditions, HIV and gender affirmation care pathways of transgender people living with HIV in France: a nationwide, comprehensive, cross-sectional, community-based research protocol (ANRS Trans&HIV). BMJ Open. 2021 Dec 16;11(12):e052691. doi: 10.1136/bmjopen-2021-052691. PMID 34916316